CLINICAL TRIAL: NCT05012735
Title: An Evaluation of the Safety and Efficacy of a Hydrocolloid Bandage on Pimples
Brief Title: A Study of a Hydrocolloid Bandage on Pimples
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCSTOH003710; CCSTOH003710 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2021-07-19; First posted 2021-08-19 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Group: Prototype Ultrathin Hydrocolloid Bandage and Study Cleanser (Experimental): Participants will wash their faces with the study cleanser (Neutrogena Ultra Gentle Daily Cleanser with Pro Vitamin B5) in the evening prior to bandage application and in the morning after removing the bandage(s) on Days 0 through 7. On Days 7 through 14, no bandages will be worn and participants will wash their faces with the study cleanser (Neutrogena Ultra Gentle Daily Cleanser with Pro Vitamin B5) in the morning and evening. Participants will cover their closed and popped pimples in the evening with 1 or 2 bandages on Days 0 through 6.
  Interventions: Drug: Study Cleanser (Neutrogena Ultra Gentle Daily Cleanser with Pro Vitamin B5); Device: Prototype Ultrathin Hydrocolloid Bandage
- Control Group: Study Cleanser (Neutrogena Ultra Gentle Daily Cleanser with Pro Vitamin B5) (Active Comparator): Participants will wash their face twice daily using the study cleanser (Neutrogena Ultra Gentle Daily Cleanser with Pro Vitamin B5) for up to 14 days.
  Interventions: Drug: Study Cleanser (Neutrogena Ultra Gentle Daily Cleanser with Pro Vitamin B5)

INTERVENTIONS:
Drug: Study Cleanser (Neutrogena Ultra Gentle Daily Cleanser with Pro Vitamin B5) — Participants will wash their face with the study cleanser (Neutrogena Ultra Gentle Daily Cleanser with Pro Vitamin B5) for up to 14 days.
Device: Prototype Ultrathin Hydrocolloid Bandage — Participants will cover their closed and popped pimples in the evening with one or two bandages from Days 0 through 6.
  Arms: Treatment Group: Prototype Ultrathin Hydrocolloid Bandage and Study Cleanser

SUMMARY:
The purpose of this study is to evaluate the effectiveness and tolerability of a hydrocolloid bandage on pimples when used overnight for one week.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and follow the requirements and restrictions of the study (including willingness to use the assigned study products per instructions, refrain from excessive sunlight and tanning booths/beds, stop all other acne product usage; availability on scheduled visit dates and likeliness of completing the clinical study) based upon research site personnel's assessment
* Evidence of a personally signed and dated informed consent or parent/guardian signed and dated informed consent (and/or assent, as applicable) document, Consent for Photograph/Video Release, including Health Insurance Portability and Accountability Act (HIPAA) disclosure, indicating the participant (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* Fitzpatrick Skin Type I to VI
* Generally in good health based on medical history
* Able to read, write, speak, and understand English
* Willing to tell the study staff or principal investigator (PI) about any health problems or new medications that they may start taking during the study
* Must have at least 1 identifiable target inflammatory/closed lesion in the active stage (between 2.0 and 5.0 millimeters [mm] in diameter)
* Must have at least 1 mature inflammatory (to-be-popped) acne lesion (papule or pustule, at least 3 mm in diameter, and capable of being extracted)

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skincare products, adhesive bandages, latex, wound treatment products, or ingredients in the investigational study materials
* Presents with a skin condition that may influence the outcome of the study, increase risk to the participant, or interfere with study evaluations, in the opinion of the PI (example., severe acne, acne conglobata, psoriasis, atopic dermatitis, eczema, cutaneous xerosis, erythema, active skin cancer, skin dermatoses, keloids, hypertrophic scars, cracked/excoriated skin, pigmentation, friable skin, or clinically infected skin lesions)
* Per Investigator's Global Assessment (IGA) of acne severity score greater than (>) 3 (moderate) according to scale where 0=Clear and 5=Very Severe
* Has a known history of severe systemic immune system disorders
* Has a known history of severe systemic immune system disorders or uncontrolled chronic diseases (such as hypertension, hyperthyroidism, hypothyroidism, or skin cancer within past year)
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication
* Is taking medications that would mask an adverse event (AE) or influence the study results, including a) antibiotics, anti-coagulants, antiplatelet drugs, cytotoxic agents, continuous aspirin therapy, chemotherapy, or daily medications for chronic asthma within 1 month before Visit 1; b) immunosuppressive drugs and steroidal and/or non-steroidal anti-inflammatory drugs within 3 months before Visit 1 and during the study; c) antihistamines within 1 month before Visit 1 and during the study
* Is self-reported to be breastfeeding, pregnant or planning to become pregnant during the study
* Has taken/used (oral or topical) vitamin A derivatives such as accutane, isotretinoin, or retinoic acid within 6 months
* Currently taking, of have taken or used on the test area any of the following in the indicated time frame before study enrollment: a) oral or topical prescription medications for acne such as azelaic acid, benzoyl peroxide, Bactrim, clindamycin, dapsone, differin, doxycycline, drospirenone, Epiduo, erythromycin, minocycline, sodium sulfacetamide, spironolactone, tetracycline, and topical tretinoin (adapalene, retin A, renova, tazarotene), vibramycin, within 30 days; b) any systemic medication considered to affect the course of acne, specifically, but not exclusively, antibiotics or steroids, within 30 days. Any topical over-the-counter (OTC) acne products (example, benzoyl peroxide, salicylic acid, and/or alpha/beta/poly-hydroxy products or medicated cleansers, wipes, masks, scrubs, gels and creams) or any facial treatment products containing retinol, retinaldehyde, retinyl esters, salicylic acid, and/or alpha/beta/poly-hydroxy products within 4 weeks
* Has a history of or a concurrent health condition/situation which, in the opinion of the PI or study physician may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Is simultaneously participating in any other clinical study or has participate in another clinical study in the past 4 weeks
* Is an employee/contractor or immediate family member of the PI, study site, or sponsor
* Has observable suntan, scars, nevi, tattoo, excessive hair (including beard, mustache, or goatee), or other dermal conditions on the face that that could interfere with study evaluations or confound study results, as determined by the PI or designee
* Coronavirus Disease 2019 (COVID-19): a) history of a confirmed COVID-19 infection in the last 30 days; b) contact with COVID-19-infected person within 14 days prior to enrollment; c) any international travel within 14 days prior to enrollment including members in the same household; d) participants with self-reported COVID-19 symptoms within the past 2 weeks: i) unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomach aches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, fever, or chest pain/tightness; ii) temperature greater than or equal to (>=) 38.0 degree Celsius (°C) /100.4° Fahrenheit (F), measured by thermometer which is adjusted for core temperature; iii) use of fever or pain reducers within the past 2 days of each onsite visit

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in General Wound Appearance Score of the Popped Pimple | Baseline (Day 0) up to Day 14
  Change from baseline in general wound appearance of the popped pimple will be assessed. It is evaluated on a scale from 0 to 4 with 0=poor (new or fresh wound with the epithelium layer missing, wound bed appears raw and possibly oozing); 1=fair (epithelial growth is starting to occur, wound bed is dry); 2=good (epithelial growth is clearly evident, wound bed color is no more than moderate erythema, scabbing may be present); 3=very good (wound bed indentation is slightly visible, wound area is mostly covered with epithelial regrowth, slight scabbing may be present); 4=excellent (fully healed, skin flush against surrounding skin, slight color mismatch may be present), with higher scores indicating a better outcome.
Percentage of Healed Popped Pimples | Baseline (Day 0) up to Day 14
  Percentage of healed popped pimples is defined as general wound appearance score greater than or equal to (>=) 3.5. General wound appearance is evaluated on a scale from 0 to 4 with 0=poor (new or fresh wound with the epithelium layer missing, wound bed appears raw and possibly oozing); 1=fair (epithelial growth is starting to occur, wound bed is dry); 2=good (epithelial growth is clearly evident, wound bed color is no more than moderate erythema, scabbing may be present); 3=very good (wound bed indentation is slightly visible, wound area is mostly covered with epithelial regrowth, slight scabbing may be present); 4=excellent (fully healed, skin flush against surrounding skin, slight color mismatch may be present), with higher scores indicating a better outcome.
Change from Baseline in Full Face Cutaneous Tolerance as Assessed by Trained Graders | Baseline (Day 0) up to Day 14
  Change from baseline in full face cutaneous tolerance as assessed by trained graders will be reported. It is evaluated on 3 criteria's: erythema, edema and dryness/scaling, all with a range of 0=none/absent, 1=mild, 2=moderate, and 3=severe, with higher scores indicating a worse outcome.
Change from Baseline in Full Face Cutaneous Tolerance as Assessed by Participants | Baseline (Day 0) up to Day 14
  Change from baseline in full face cutaneous tolerance as assessed by participants will be reported. It is evaluated on 3 criteria's: burning/stinging, itching and tight/dry feeling, all with a range of 0=none (no burning/stinging or itching or no skin tightness/dry feeling of the treatment area); 1= mild (slight burning/stinging sensation or itching or definite tightness or dry feeling of the treatment area; not really bothersome); 2=moderate (definite warm burning/stinging or itching or tightness or dry feeling of the treatment area that is somewhat bothersome) 3=severe (marked burning/stinging sensation or itching sensation or tightness/dry feeling of the treatment area that causes definite discomfort and may interrupt daily activities and/or sleep), with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Change from Baseline in Clinical Grading of Wound Healing of Edema of a Popped Pimple | Baseline (Day 0) up to Day 14
  Change from baseline in clinical grading of wound healing of a popped pimple will be reported. Grading of edema will be evaluated on a scale of 0 to 4 with 0=none/absent, 1=mild, 2=moderate, 3=marked; and 4=severe, with higher scores indicating a worse outcome.
Change from Baseline in Clinical Grading of Wound Healing of Crusting/Scabbing of a Popped Pimple | Baseline (Day 0) up to Day 14
  Change from baseline in clinical grading of wound healing of crusting/scabbing of a popped pimple will be reported. Grading of crusting/scabbing will be evaluated on a scale of 0 to 4 with 0=none; 1=slight (up to 30 percent [%]); 2=moderate (31% to 60%); 3=extensive (61% to 90%); and 4=almost complete or complete (91% to 100%), with higher scores indicating a worse outcome.
Change from Baseline in Clinical Grading of Wound Healing of Smoothness of a Popped Pimple | Baseline (Day 0) up to Day 14
  Change from baseline in clinical grading of wound healing of smoothness of popped pimple as assessed by trained grader will be reported. Grading of smoothness will be evaluated on a scale of 0 to 4 with 0=rough, uneven wound, 1=mild smoothness, 2=moderate smoothness, 3=extensive smoothness, and 4=complete smooth, even wound, with higher scores indicating a better outcome.
Change from Baseline in Clinical Acne Grading of Erythema of a Closed and Popped Pimples | Baseline (Day 0) up to Day 14
  Change from baseline in clinical acne grading of erythema of a closed and popped pimple will be reported. Grading of erythema will be evaluated on a scale of 0 to 4 with 0=none, 1=slight, 2=mild, 3=moderate, and 4=severe, with higher scores indicating a worse outcome.
Change from Baseline in Clinical Acne Grading of Size (Diameter) of a Closed and Popped Pimples | Baseline (Day 0) up to Day 14
  Change from baseline in clinical acne grading of size (diameter) of a closed and popped pimple will be reported. Grading of size will be evaluated on a scale of 0 to 4 with 0=no visible lesion, 1=slightly visible lesion; less than (<) 2 millimeters (mm), 2=small lesion; 2.0 mm to 3.0 mm, 3=medium lesion; 3.1 mm to < 5.0 mm, and 4=large lesion; greater than or equal to (>=) 5.0 mm, with higher scores indicating a worse outcome.
Change from Baseline in Clinical Acne Grading of Elevation of a Closed and Popped Pimples | Baseline (Day 0) up to Day 14
  Change from baseline in clinical acne grading of elevation of a closed and popped pimple will be reported. Grading of elevation will be evaluated on a scale of 0 to 4 with 0=completely flat, 1=slightly raised, 2=mildly raised, 3=moderately raised, and 4=severely raised, with higher scores indicating a worse outcome.
Change from Baseline in Clinical Acne Grading of Dryness/Scaling of a Closed and Popped Pimples | Baseline (Day 0) up to Day 14
  Change from baseline in clinical acne grading of dryness/scaling of a closed and popped pimple will be reported. Grading of dryness/scaling will be evaluated on a scale of 0 to 4 with 0=none, 1=mild, 2=moderate, and 3=severe, with higher scores indicating a worse outcome.
Change from Baseline in Investigator's Global Assessment (IGA) of Acne Severity | Baseline (Day 0) up to Day 14
  Change from baseline in IGA of acne severity will be reported. The IGA scale for acne reflects the Investigator's assessment of the severity of a participant's acne on a scale from 0 to 5 with 0 (clear skin), 1 (almost clear), 2 (mild), 3 (moderate), 4 (severe), 5 (very severe). Each of these gradations is based upon a lesion count by the Investigator.
Microbiome Analysis of Closed and Popped Pimple | Baseline (Day 0) and Day 7
  Microbiome analysis of closed and popped pimple for Days 0 and 7 will be reported. Microbiome sample swabs will be used to collect bacteria from the skin surface and will be processed by CosmosID Inc using spike-in quantification controls and shallow shotgun metagenome sequencing at 3-4 millions (M) reads per sample.
Consumer Perception Questionnaire | Up to Day 13
  Consumer perception will be assessed quantitatively by consumer perception questionnaire which consists of some questions regarding how participants feel about using the bandages. In order to capture this information, a smartphone app called dscout will be used that will allow the participants to easily provide the information with a glimpse of the experience. In each research activity, participants will be asked to answer a set of questions and submit a photo and/or video of him/her.
Standardized Digital Photographs of Full Face | Baseline (Day 0) up to Day 14
  Standardized digital photographs of full face (right, center, left) will be captured using the Johnson & Johnson (J&J) Lab Imaging System for qualitative image analysis. It will assess visual improvements in closed and popped pimples.

CONTACTS AND LOCATIONS:
Overall Officials: Summer Acevedo, PhD, Principal Investigator — Stephens SGS, Inc.
Locations (1):
- SGS Stephens Inc., Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Heng AHS, Chew FT. Systematic review of the epidemiology of acne vulgaris. Sci Rep. 2020 Apr 1;10(1):5754. doi: 10.1038/s41598-020-62715-3. PMID 32238884
- [Background] Tripathi SV, Gustafson CJ, Huang KE, Feldman SR. Side effects of common acne treatments. Expert Opin Drug Saf. 2013 Jan;12(1):39-51. doi: 10.1517/14740338.2013.740456. Epub 2012 Nov 20. PMID 23163336
- [Background] Mayo Foundation for Medical Education and Research. Acne Treatment. Retrieved from https://www.mayoclinic.org/diseases-conditions/acne/diagnosis-treatment/drc-20368048
- [Background] Chao CM, Lai WY, Wu BY, Chang HC, Huang WS, Chen YF. A pilot study on efficacy treatment of acne vulgaris using a new method: results of a randomized double-blind trial with Acne Dressing. J Cosmet Sci. 2006 Mar-Apr;57(2):95-105. PMID 16688374
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSTOH003710&attachmentIdentifier=bc101dd9-e7c2-46b3-abc8-34a86c8f7ae8&fileName=CCSTOH003710_CSR_Synopsis_for_Posting.pdf&versionIdentifier=